CLINICAL TRIAL: NCT03238183
Title: Additional Therapeutic Effects of Dextrose to Hyaluronic Acid on Knee Osteoarthritis: a Double Blind, Randomized-controlled Clinical Trial
Brief Title: Effects of Dextrose on Knee Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOST 106-2314-B-341-003
Record Dates: First submitted 2017-07-28; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Physical Activity; Functional Disturbance
Keywords: knee osteoarthritis; hyaluronic acid; dextrose; therapeutic effects
MeSH Terms: conditions — Motor Activity; Osteoarthritis, Knee | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyaluronic acid combined dextrose group (Active Comparator): Hyaluronic acid (2 cc) combined 25% dextrose (3.5 cc 50% dextrose plus 3.5 cc 2% lidocaine) injection: one injection per week, for 3 weeks, to compare the additional therapeutic effects of combined hyaluronic acid and dextrose injections to hyaluronic acid injections
  Interventions: Drug: dextrose; Device: hyaluronic acid
- hyaluronic acid group (Placebo Comparator): Hyaluronic acid (2 cc) combined normal saline (3.5 cc normal saline plus 3.5 cc 2% lidocaine) injection: one injection per week, for 3 weeks, to compare the additional therapeutic effects of combined hyaluronic acid and dextrose injections to hyaluronic acid injections
  Interventions: Device: hyaluronic acid

INTERVENTIONS:
Drug: dextrose — compare the therapeutic effects of hyaluronic acid combined dextrose injections with hyaluronic acid injections only to patients with knee osteoarthritis
  Other Names: glucose water
  Arms: hyaluronic acid combined dextrose group
Device: hyaluronic acid — compare the therapeutic effects of hyaluronic acid combined dextrose injections with hyaluronic acid injections only to patients with knee osteoarthritis

SUMMARY:
Using double blind, randomized controlled design to study the immediate, short-term and intermediate-term therapeutic effects of ultrasound guided hyaluronic acid injection and hyaluronic acid combined dextrose injection to patients with knee osteoarthritis.

DETAILED DESCRIPTION:
A total of 106 patients will be collected. The participants will be randomized into two groups, including hyaluronic acid group and hyaluronic acid combined dextrose group.

The hyaluronic acid group will receive 3 times of hyaluronic acid injection per week in three weeks; the hyaluronic acid combined dextrose group will receive 3 times of hyaluronic acid combined dextrose injection per week in three weeks.

The pain, physical activity, and functional performance will be evaluated.

All the evaluations will be re-evaluated at one week after injection, one month after injection, three months after injection, and six month after injection.

Subjects and the evaluator will be both blinded to the group's classification during the whole course of study.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis with Kellgren/Lawrence grade II or III

Exclusion Criteria:

* who have neurological deficit, such as stroke who have implant in knee

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
physical activity-on level walking time | changes from baseline to at one week after injection, one month after injection, three months after injection, and six month after injection
  10 meter walking
physical activity-stair climbing time | changes from baseline to at one week after injection, one month after injection, three months after injection, and six month after injection
  stairs climbing
physical activity-chair rising time | changes from baseline to at one week after injection, one month after injection, three months after injection, and six month after injection
  chair rising

SECONDARY OUTCOMES:
functional performance | changes from baseline to at one week after injection, one month after injection, three months after injection, and six month after injection
  Western Ontario and McMaster Universities Osteoarthritis index
quality of life | changes from baseline to at one week after injection, one month after injection, three months after injection, and six month after injection
  Knee Injury and Osteoarthritis Outcome Score

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsieh RL, Lee WC. Effects of Intra-articular Coinjections of Hyaluronic Acid and Hypertonic Dextrose on Knee Osteoarthritis: A Prospective, Randomized, Double-Blind Trial. Arch Phys Med Rehabil. 2022 Aug;103(8):1505-1514. doi: 10.1016/j.apmr.2022.04.001. Epub 2022 Apr 16. PMID 35439521